CLINICAL TRIAL: NCT01096966
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Efficacy and Safety of Bupivacaine TTS (Bupivacaine Patch) in Patients With Chronic Low Back Pain
Brief Title: Study of the Efficacy and Safety of Bupivacaine TTS Patch in Patients With Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durect (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K843-09-2001
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine TTS (Experimental)
  Interventions: Drug: Bupivacaine TTS (Bupivacaine Patch)
- Placebo patch (Placebo Comparator)
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: Bupivacaine TTS (Bupivacaine Patch) — Contains bupivacaine base, in a flexible and rectangular-shaped, transdermal, delivery system. Three patches applied to the lower back every 72 hours for 12 weeks.
  Arms: Bupivacaine TTS
Drug: Placebo patch — Identical in size and shape to the Bupivacaine Patch. Three patches applied to the lower back every 72 hours for 12 weeks.
  Arms: Placebo patch

SUMMARY:
This study will evaluate the efficacy and safety of Bupivacaine TTS (Bupivacaine patch) compared to placebo in patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic low back pain for more than 3 months
2. If taking non-steroidal anti-inflammatory drugs or non-opioid analgesics, must be on a regular, scheduled dose for at least 4 weeks prior to the first visit and intend to remain on a stable dose of these agents for the study duration
3. Pain intensity score greater than or equal to 5 out of 10 at the first visit
4. Able to apply patches at home
5. Able and willing to complete daily pain intensity ratings using an electronic diary device for the duration of the study
6. Females of childbearing potential must agree to use a medically acceptable method of contraception throughout the study

Exclusion Criteria:

1. History of, or ongoing, alcohol or drug abuse
2. Positive drug test for alcohol, illicit drug use or opioids
3. Primary diagnosis of chronic low back pain due to neuropathic pain
4. History of back surgery or plan for back surgery
5. Use of opioids within 2 weeks of the first visit and during the study
6. Previous ineffective use of lidocaine patches
7. Morbid obesity
8. Moderate or severe depression
9. An open skin lesion within the painful area where patches will be applied
10. Patients with active or resolved back pain litigation or receiving disability payments due to chronic low back pain
11. Pregnant or breastfeeding females

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to 12 weeks in pain in the last 24 hours (daily scores averaged over 14 days) | baseline to 12 weeks after baseline

SECONDARY OUTCOMES:
Subjects achieving 20% pain relief at 12 weeks compared to baseline | baseline to 12 weeks after baseline
Subjects 'much improved' or 'very much improved' at 12 weeks | 12 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul Meisner, PharmD, Study Director — King Pharmaceuticals is now a wholly owned subsidiary of Pfizer
Locations (21):
- United States (21):
  - Tempe, Arizona
  - La Mesa, California
  - Torrance, California
  - Fort Lauderdale, Florida
  - Gainesville, Florida
  - Longwood, Florida
  - West Palm Beach, Florida
  - Marietta, Georgia
  - Newnan, Georgia
  - Springfield, Massachusetts
  - St Louis, Missouri
  - New York, New York
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Altoona, Pennsylvania
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Richmond, Virginia